CLINICAL TRIAL: NCT04320264
Title: Metabolic Inflexibility is Related to Elevated Muscle Anaerobic Glycolysis
Status: Recruiting | Type: Observational
Sponsor: East Carolina University (Other)
Collaborators: Duke University (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: UMCIRB 19-000914
Record Dates: First submitted 2019-09-03; First posted 2020-03-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Inflexibility
Keywords: Metabolic Inflexibility; Obesity; Anaerobic glycolysis
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and tissue samples without analysis of DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low oxidizers/high lactate: Individuals with low aerobic oxidation
- High oxidizers/low lactate: Individuals with high aerobic oxidation
- Obese: Severely obese scheduled for surgery
  Interventions: Procedure: Weight loss surgery

INTERVENTIONS:
Procedure: Weight loss surgery — Severely obese women (BMI >40) undergo sleeve gastrectomy
  Groups: Obese

SUMMARY:
The focus of this proposal is on overweight (25>BMI<30 kg/m2) subjects, as these individuals exhibit a high risk of becoming obese and/or developing metabolic diseases. We hypothesize that in some overweight individuals there is a "metabolic program" in skeletal muscle which predisposes them to the development of obesity. Findings may lead to clinical screening tools for determining risk for obesity in non-obese individuals and targeting this group for prevention.

DETAILED DESCRIPTION:
Our overall hypothesis is that increased reliance on anaerobic glycolysis in muscle shifts fasting metabolism from fat towards carbohydrate utilization, which results in metabolic inflexibility and subsequent metabolic disease (i.e. obesity). To test our hypothesis, overweight subjects (BMI 25 to 30 kg/m2) will be recruited and screened for reliance on anaerobic glycolysis (resting/fasting plasma lactate concentrations). Subjects with high (top quartile) and low (bottom quartile) resting/fasting plasma lactate will be chosen. The premise of this screening is that subjects with low lactate will have high muscle aerobic substrate oxidation, while those with elevated lactate will have low muscle oxidative metabolism. Severely obese subjects will be studied as a comparator group. In aim 1 in vivo muscle lactate release and respiratory exchange ratio (RER) will be determined to investigate if subjects with high reliance on anaerobic glycolysis exhibit a shift towards carbohydrate utilization at the whole-body level. Aim 2 will test whether subjects with elevated reliance on anaerobic glycolysis in muscle are metabolically inflexible. To establish causality, aim 3 is designed to follow subjects after an intervention that shifts skeletal muscle metabolism from carbohydrate to fat utilization. Our preliminary findings indicate that bariatric surgery normalizes muscle lactate production; therefore, severely obese subjects will be studied before and after gastric bypass surgery (aim 3).

The study (MetFlex) will enroll 74 adults; (Group 1) 60 overweight (BMI 25 to 30 kg/m2) males and females ages 18-50 years old and (Group 2) 14 severely obese (BMI 40 to 50 kg/m2) adult females who are scheduled for bariatric surgery.

Endpoints to be investigated in the 3 specific aims.

Carbohydrate/fat oxidation (RER) in the fasting condition. High lactate vs low lactate groups (aim 1). Pre-surgery vs post-surgery (aim 3)

Muscle oxygen consumption (substrate oxidation) in the fasting condition. High lactate vs low lactate groups (aim 1). Pre-surgery vs post-surgery (aim 3)

Muscle lactate release in the fasting condition. High lactate vs low lactate groups (aim 1). Pre-surgery vs post-surgery (aim 3)

Endogenous glucose production in the fasting condition. High lactate vs low lactate groups (aim 1). Pre-surgery vs post-surgery (aim 3)

Insulin sensitivity (clamp M value). High lactate vs low lactate groups (aim 1)

Change in Carbohydrate/fat oxidation (RER) in response to glucose + insulin (metabolic flexibility). High lactate vs low lactate groups (aim 2)

Change in muscle fat oxidation in response to high fat feeding (metabolic flexibility). High lactate vs low lactate groups (aim 2)

Change in muscle oxygen consumption (substrate oxidation) in response to high fat feeding (metabolic flexibility). High lactate vs low lactate groups (aim 2)

Our basic premise is that elevated fasting plasma lactate causes glucose production to be increased and that a "Vicious Cori cycle" is the underlying cause of the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* BMI of 25 - 30 kg/m2
* BMI > 40kg/m2
* Lactate levels in top and lower 25%

Exclusion Criteria:

* Pregnant women
* Mentally disabled
* Prisoners
* Smokers
* Subjects with heart disease
* Type 1 and 2 diabetes
* Endocrine disease
* Hypertension
* Musculoskeletal disease
* Peripheral occlusion
* Hepatic disease
* Have had weight fluctuations exceeding + 3% in the previous 12 months
* On medications which alter carbohydrate metabolism will not be studied

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: High oxidizers Low oxidizers Obese
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Carbohydrate/fat oxidation (RER) in the fasting condition. | Years 1-5
  RER will be measured from indirect calorimetry
Muscle oxygen consumption (substrate oxidation) in the fasting condition. | Years 1-5
  Muscle oxygen consumption will be measured by near-infrared spectroscopy (NIRS)
Muscle lactate release in the fasting condition. | Years 1-5
  Muscle lactate release will be measured by microdialysis
Change in Carbohydrate/fat oxidation (RER) in response to glucose + insulin (metabolic flexibility) | Years 1-5
  Indirect calorimetry during glucose clamp
Change in muscle fat oxidation in response to high fat feeding (metabolic flexibility). | Years 1-5
  Oxidation of fatty acid in muscle homogenate.
Change in muscle oxygen consumption (substrate oxidation) in response to high fat feeding (metabolic flexibility). | Years 1-5
  Oxygen consumption measured by near-infrared spectroscopy (NIRS)

SECONDARY OUTCOMES:
Insulin sensitivity (clamp M value). | Years 1-5
  Measured during glucose clamp.
Endogenous glucose production in the fasting condition. | Years 1-5
  Measured with isotopically labeled glucose

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Houmard, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan TE, Brophy P, Lin CT, Hickner RC, Neufer PD. Assessment of in vivo skeletal muscle mitochondrial respiratory capacity in humans by near-infrared spectroscopy: a comparison with in situ measurements. J Physiol. 2014 Aug 1;592(15):3231-41. doi: 10.1113/jphysiol.2014.274456. Epub 2014 Jun 20. PMID 24951618
- [Background] Camisa C, Rossana C. Variant of keratoderma hereditaria mutilans (Vohwinkel's syndrome). Treatment with orally administered isotretinoin. Arch Dermatol. 1984 Oct;120(10):1323-8. PMID 6237617
- [Background] Craglietto T, Giarelli L, Paolini A. [Comparative study of the DNA content of human female breast adenocarcinomas and of their recurrences. (Histo-spectrophotometric findings)]. Riv Anat Patol Oncol. 1964 Nov-Dec;26(5):694-706. No abstract available. Italian. PMID 5866193
- [Background] Ciresa M, Gabl F, Knapp E. [Acid-base equilibrium]. Wien Klin Wochenschr. 1970 Jan 2;82(1):11-2. No abstract available. German. PMID 5513193
- [Background] Iwamasa J, Tajima C, Matsuura K, Okamura H. [Role of progesterone in the ovulatory process of PMSG/hCG treated immature female rats]. Nihon Sanka Fujinka Gakkai Zasshi. 1989 Oct;41(10):1551-6. Japanese. PMID 2584808